CLINICAL TRIAL: NCT01084603
Title: Single-dose Nicotine Pharmacokinetics With a New Oral Nicotine Replacement Product. A Study in Healthy Smokers
Brief Title: Single-dose Nicotine Pharmacokinetics With a New Oral Nicotine Replacement Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NICTDP1065/A6431116; 2008-006280-36 (EudraCT Number)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2010-07-08 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Oral Nicotine 1 (Experimental): One oral administration of 1 mg nicotine
  Interventions: Drug: Oral Nicotine
- Oral Nicotine 2 (Experimental): Two oral administrations of 1 mg nicotine
  Interventions: Drug: Oral Nicotine
- Oral Nicotine 4 (Experimental): Four oral administrations of 1 mg nicotine
  Interventions: Drug: Oral Nicotine
- NiQuitinTM Nicotine Lozenge 4 mg (Active Comparator): One 4 mg marketed nicotine lozenge
  Interventions: Drug: NiQuitinTM Nicotine Lozenge
- Nicorette® Gum 4 mg (Active Comparator): One marketed Nicorette® nicotine gum 4 mg chewed for 30 minutes
  Interventions: Drug: Nicorette® Nicotine Gum

INTERVENTIONS:
Drug: Oral Nicotine — A new l mg oral nicotine product
  Other Names: Experimental nicotine 1 mg
  Arms: Oral Nicotine 1; Oral Nicotine 2; Oral Nicotine 4
Drug: NiQuitinTM Nicotine Lozenge — A marketed 4 mg Nicotine lozenge
  Other Names: NiQuitinTM lozenge
  Arms: NiQuitinTM Nicotine Lozenge 4 mg
Drug: Nicorette® Nicotine Gum — A marketed 4 mg Nicotine Gum
  Other Names: Nicorette® gum
  Arms: Nicorette® Gum 4 mg

SUMMARY:
A comparison of three products for oral nicotine replacement with respect to pharmacokinetics after single-dose of nicotine.

DETAILED DESCRIPTION:
This study compares a new oral Nicotine Replacement Therapy (NRT) product with NiQuitin™ lozenge 4 mg and Nicorette®gum 4 mg, after 12 hours of nicotine abstinence, with respect to nicotine pharmacokinetics, during 12 hours after start of administration. Single doses of each treatment are given once in the morning during five separate treatment visits scheduled in a crossover setting with randomized treatment sequences. The study will include 45 healthy smokers between 18-50 years, who have been smoking at least 15 cigarettes daily during at least one year preceding inclusion. Subjects and study personnel will be aware of which treatment is administered at a given visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy smokers, smoking at least 15 cigarettes daily during at least one year preceding inclusion and BMI between 17.5 and 30.0 kg/m2.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 months preceding the first dose of study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Clinical Pharmacology, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Full Safety Set
Period: Baseline
Arm/Group | Overall Study
Started | 45
Completed | 43
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: NiQuitinTM Lozenge
Arm/Group | Overall Study
Started | 43
Completed | 42
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Washout Period 1
Arm/Group | Overall Study
Started | 42
Completed | 42
Not Completed | 0
Period: Nicorette® Gum
Arm/Group | Overall Study
Started | 42
Completed | 41
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Washout Period 2
Arm/Group | Overall Study
Started | 41
Completed | 41
Not Completed | 0
Period: Oral Nicotine 1
Arm/Group | Overall Study
Started | 41
Completed | 40
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Washout Period 3
Arm/Group | Overall Study
Started | 40
Completed | 40
Not Completed | 0
Period: Oral Nicotine 2
Arm/Group | Overall Study
Started | 40
Completed | 40
Not Completed | 0
Period: Washout Period 4
Arm/Group | Overall Study
Started | 40
Completed | 39
Not Completed | 1
Not completed — Adverse Event | 1
Period: Oral Nicotine 4
Arm/Group | Overall Study
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 24
Region of Enrollment [Number; unit: participants]
  Sweden | 45

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration
Description: Cmax, which is the maximum (peak) concentration (amount of drug) measurable in blood plasma after a dose is administered measured in nanograms/milliliter (ng/ml)
Time Frame: During 12 hours after start of administration
Population: ITT
Measure: Geometric Mean (Standard Deviation); unit: (ng/ml)
Groups:
- Oral Nicotine 1: 1 administration of 1 mg
- Oral Nicotine 2: 2 administrations of 1 mg
- Oral Nicotine 4: 4 administrations of 1 mg
- NiQuitinTM Lozenge 4 mg: 1 NiQuitinTM nicotine lozenge 4 mg
Arm/Group | Oral Nicotine 1 | Oral Nicotine 2 | Oral Nicotine 4 | NiQuitinTM Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 40 | 40 | 39 | 42 | 41
(ng/ml) | 3.04 (1.47) | 4.94 (2.06) | 8.63 (2.96) | 6.44 (2.06) | 7.36 (2.66)

2. Secondary Outcome: Nicotine Plasma Concentration
Description: Area under the nicotine plasma concentration curve at 10 minutes (AUC10 min)
Time Frame: During 10 minutes after start of administration
Population: ITT
Measure: Geometric Mean (Standard Deviation); unit: (h*ng/ml)
Arm/Group | Oral Nicotine 1 | Oral Nicotine 2 | Oral Nicotine 4 | NiQuitinTM Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 40 | 40 | 39 | 42 | 41
(h*ng/ml) | 0.43 (0.23) | 0.56 (0.33) | 0.87 (0.42) | 0.29 (0.20) | 0.29 (0.20)

3. Secondary Outcome: Time of Maximum Concentration
Description: The time at which maximum concentration is reached (Tmax)
Time Frame: During 12 hours after start of administration
Population: ITT
Measure: Median (Full Range); unit: (hours)
Arm/Group | Oral Nicotine 1 | Oral Nicotine 2 | Oral Nicotine 4 | NiQuitinTM Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 40 | 40 | 39 | 42 | 41
(hours) | 0.17 [0.07 to 1.50] | 0.21 [0.07 to 1.00] | 0.17 [0.07 to 1.50] | 0.75 [0.17 to 2.02] | 0.50 [0.33 to 1.00]

4. Secondary Outcome: Terminal Elimination Rate Constant
Description: The terminal nicotine elimination rate constant (Lamda z)
Time Frame: During 12 hours after start of administration
Population: ITT
Measure: Mean (Standard Deviation); unit: (1/hr)
Arm/Group | Oral Nicotine 1 | Oral Nicotine 2 | Oral Nicotine 4 | NiQuitinTM Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 40 | 40 | 39 | 42 | 41
(1/hr) | 0.29 (0.13) | 0.29 (0.10) | 0.30 (0.10) | 0.26 (0.07) | 0.31 (0.10)

5. Secondary Outcome: Released Nicotine
Description: The amount of nicotine released from Nicorette® gum 4 mg during 30 minutes' chewing
Time Frame: After 30 minutes' chewing
Population: ITT
Measure: Mean (Standard Deviation); unit: (ng/ml)
Arm/Group | Nicorette® Gum 4 mg
Number analyzed (Participants) | 41
(ng/ml) | 2.70 (0.27)

6. Primary Outcome: Bioavailability
Description: A measure of how much of the drug reaches a person's bloodstream within a given period of time for the body to use. The extent of product bioavailability is estimated by the area under the blood concentration vs time curve. The area under the curve (AUC) is calculated by plotting the drug's blood levels on a graph at different times during the set period to form a curve. The area under this curve reflects the amount of drug exposure in the set time period, calculated as hour*nanograms/milliliter (h*ng/ml).
Time Frame: 12 hours
Measure: Geometric Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Oral Nicotine 1 | Oral Nicotine 2 | Oral Nicotine 4 | NiQuitinTM Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 40 | 40 | 39 | 42 | 41
h*ng/ml
  AUC to last measurable concentration | 5.85 (3.7) | 11.50 (3.98) | 21.96 (9.00) | 22.00 (11.05) | 19.69 (7.95)
  AUC to infinity | 7.54 (4.10) | 13.30 (4.20) | 24.10 (9.35) | 24.30 (11.91) | 21.62 (8.43)

ADVERSE EVENTS:
Arm/Group | Oral Nicotine 1 | Oral Nicotine 2 | Oral Nicotine 4 | NiQuitinTM Lozenge 4 mg | Nicorette® Gum 4 mg
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/42 | 0/43 | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 11/41 | 11/42 | 24/43 | 7/43 | 9/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Nicotine 1 (N=41) | Oral Nicotine 2 (N=42) | Oral Nicotine 4 (N=43) | NiQuitinTM Lozenge 4 mg (N=43) | Nicorette® Gum 4 mg (N=42)
Appendicitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Nicotine 1 (N=41) | Oral Nicotine 2 (N=42) | Oral Nicotine 4 (N=43) | NiQuitinTM Lozenge 4 mg (N=43) | Nicorette® Gum 4 mg (N=42)
Nausea (Gastrointestinal disorders) | 2 | 3 | 4 | 2 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 3 | 2 | 1
Headache (Nervous system disorders) | 7 | 1 | 6 | 5 | 4
Hiccups (Gastrointestinal disorders) | 2 | 1 | 10 | 0 | 3
Throat Irritation (Gastrointestinal disorders) | 2 | 4 | 6 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes